CLINICAL TRIAL: NCT05891418
Title: Effect of Email Nudges on Plan Switching and Healthcare Utilization Among Unemployment Insurance Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Office of Evaluation Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrew Feher, Research Scientist, Office of Evaluation Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 022023
Record Dates: First submitted 2023-02-14; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Health Behavior
Keywords: Affordable Care Act; randomized controlled trial; nudge; American Rescue Plan; unemployment insurance
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group with a standard eligibility notice (Experimental): Control group was assigned to receive no email outreach in June and July beyond an eligibility redetermination notice.
  Interventions: Behavioral: Standard notice of eligibility determination
- Treatment group with a standard eligibility notice and assigned two email nudges (Experimental): Assigned to receive an eligibility redetermination notice along with two informational emails about the benefits of Cost-Sharing Reduction Silver plans.
  Interventions: Behavioral: Two informational emails with plan information

INTERVENTIONS:
Behavioral: Two informational emails with plan information — Informational emails about the benefits of Cost-Sharing Reduction Silver plans.
  Arms: Treatment group with a standard eligibility notice and assigned two email nudges
Behavioral: Standard notice of eligibility determination — No extra outreach during intervention period.
  Arms: Control Group with a standard eligibility notice

SUMMARY:
In March 2021, President Biden signed into law the American Rescue Plan Act of 2021 (ARP), a landmark federal economic relief and stimulus package designed to provide support to Americans hit by the economic recession brought about by the COVID-19 global pandemic. The law provides increased federal premium tax credits (PTC), and ensures that consumers will pay no more than 8.5 percent of household income on health insurance premiums in 2021 and 2022, if enrolled through an Affordable Care Act marketplace like Covered California.

The ARP also provides additional PTC and cost-sharing reduction (CSR) benefits to eligible marketplace enrollees who report receiving unemployment insurance benefits (UIB) for at least one week in 2021. Under the law, for 2021 only, Covered California consumers will have their household income level treated as if it were at 138.1 percent of the federal poverty level (FPL), regardless of their projected annual income, which will make them eligible for a Silver 94 plan, and which offers the greatest value on cost-sharing benefits.

But in order to access those cost-sharing benefits, households must be in silver tier plans, but over 40,000 were not. This project's goal is to assess the effects of an informational email on plan switching into Cost Sharing Reduction Silver plans and downstream healthcare utilization.

The project's research design is a randomized intervention among approximately 42,500 enrolled households with an email address in non-silver tier plans. The investigators randomly assigned to either two informational emails or to a no email control group. The investigators then collected administrative data to examine plan switching behavior and healthcare utilization among households in the study.

ELIGIBILITY:
Inclusion Criteria:

* Has email address, in a non-silver plan and reported unemployment insurance in 2021

Exclusion Criteria:

* In a silver plan, no email address

Ages: 0 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42470 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Cost-Sharing Reduction Silver Enrollment | 1 month
  Percent of households enrolled in a Cost-Sharing Reduction Silver Plan
Office Visit | 6 months
  Percent of households with an office visit
Prescription drug use | 6 months
  Percent of households with a prescription drug fill
Emergency room visit | 6 months
  Percent of households with an emergency room visit
Hospitalization | 6 months
  Percent of households with a hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Feher, PhD, Principal Investigator — Covered California
Locations (1):
- Covered California, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers are committed to sharing as much data as possible for replication, consistent with the privacy and security requirements of the state agency that govern the re-disclosure of the data.
Supporting Information: Study Protocol
Time Frame: Data will be available with investigator support upon publication
Access Criteria: Replication data can be accessed via request to the primary investigator upon publication.

REFERENCES:
- [Derived] Lovchikova M, Feher A, Lian L. Health Plan Switching and Health Care Utilization: A Randomized Clinical Trial. JAMA Health Forum. 2024 Mar 1;5(3):e240324. doi: 10.1001/jamahealthforum.2024.0324. PMID 38551588

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT05891418/SAP_000.pdf